CLINICAL TRIAL: NCT00252473
Title: Evaluation of Setup Accuracy in Med Tec S-Frame Immobilization Masks For Patients Undergoing Radiation Therapy For Head and Neck Cancer
Brief Title: S-Frame CT Immobilization Masks For Patients Undergoing Radiation Therapy For Head and Neck Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: Princess Margaret Hospital, Canada (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UHN REB 02-0832-C
Record Dates: First submitted 2005-11-09; First posted 2005-11-11 (Estimated); Last update posted 2010-08-13 (Estimated); Status verified 2010-08

CONDITIONS: Head and Neck Neoplasms
MeSH Terms: conditions — Head and Neck Neoplasms

INTERVENTIONS:
Device: MedTec S-frame Immobilization Masks

SUMMARY:
Immobilization devices such as thermoplastic masks are used routinely in the radiation treatment of head and neck cancer patients. It is important to assess how well they function at preventing patient motion while the radiation treatment is being delivered. (i.e. isocentre set-up margins, patient motion with the mask). If these new thermoplastic masks such as MedTec S-frame allow less movement, then smaller margins are needed during radiation therapy which, in turn, would decrease side effects from the treatment.

ELIGIBILITY:
Inclusion Criteria:

* Histological confirmation of mucosal malignancy in the head and neck (H&N) region
* Undergoing radiotherapy (RT) with curative intent using a lateral parallel pair treatment with an anterior or anterior/posterior low neck filed technique using a MedTec S-frame mask

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2005-01; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Measurement of the accuracy of MedTec S-frame head and neck immobilization system (isocentre set-up accuracy, patient movement margins and movement of the normal tissue critical structures and planning target volumes)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Bayley, MD, Principal Investigator — Princess Margaret Hospital, Canada
Locations (1):
- University Health Network, Toronto, Ontario, Canada